CLINICAL TRIAL: NCT02391506
Title: A Prospective Study to Evaluate the Safety and Effectiveness of the Cartiva® Synthetic Cartilage Implant for CMC in the Treatment of First Carpometacarpal Joint Osteoarthritis
Brief Title: Safety and Effectiveness of Cartiva Implant in the Treatment of First CMC Joint Osteoarthritis
Acronym: GRIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cartiva, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC-0116
Record Dates: First submitted 2015-03-09; First posted 2015-03-18 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis
Keywords: First CMC joint; Osteoarthritis; Cartilage Replacement; First CMC Joint Osteoarthritis; Damaged Articular Surface
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cartiva (Experimental): Synthetic Cartilage Implant
  Interventions: Device: Cartiva

INTERVENTIONS:
Device: Cartiva — Cartiva Synthetic Cartilage Implant

SUMMARY:
This study will evaluate whether Cartiva is an effective treatment for individuals with osteoarthritis of the CMC joint in the hand.

DETAILED DESCRIPTION:
This is a prospective traditional feasibility study evaluating Cartiva® SCI for CMC for the treatment of first carpometacarpal joint osteoarthritis.The objectives of this clinical study are to evaluate the safety and effectiveness of Cartiva® SCI for CMC in terms of pain relief and improvement of joint function in the treatment of first CMC OA and to evaluate Cartiva® SCI for CMC device performance in order to establish the parameters for a pivotal trial. Follow up visits will occur at the following time points after the surgical procedure: 14 days, 42 days, 90 days, 180 days, 1 year and 2 year.

Data will be summarized using descriptive statistics. Continuous variables will be summarized using the number of observations, mean, standard deviation, median, and range as appropriate. Categorical values will be summarized using the number of observations and percentages as appropriate. Chi-square or Fisher exact tests will be used for comparisons of categorical data. Paired t-tests will used for the comparisons of continuous data. For statistical testing, an alpha of 0.05 is used as an acceptance standard and all testing are conducted as two tailed. Also, 95% confidence intervals for mean values or proportion values will be provided as appropriate.

Since this is a feasibility study and no formal hypothesis is to be tested, p-values will be reported without adjustment for multiple comparisons. All analyses will be conducted using SAS version 9.1 or later.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Osteoarthritis of the first carpometacarpal joint
* Presence of good bone stock without the need for bone graft
* Capable of completing self-administered questionnaires

Exclusion Criteria:

* < 18 years of age
* Active bacterial infection of the hand
* Previous CMC implant and/or surgery to the affected joint to be treated that would prevent implantation and fixation of Cartiva® SCI for CMC
* Patient has osteoarthritis of the scaphotrapeziotrapezoidal (STT) joint in the hand to be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Pain measured by the Visual Analog Scale (VAS) scale | 1 year follow up

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - UBC, Division of Plastic Surgery, Vancouver, British Columbia
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- United Kingdom (5):
  - Woodend Hospital, Aberdeen, Scotland
  - Royal United Hospital, Bath
  - Royal Derby Hospital, Derby
  - South Tees Hospital, Middlesbrough
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: No